CLINICAL TRIAL: NCT04145570
Title: A Single-Dose,ComparativeBioavailability Study ofTwo Formulations ofErlotinib150mgTabletsunderFastingConditions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Quadras Scientific Solutions (Other)
Responsible Party: Principal Investigator, Gastón Kuperman, Doctor Clinical - Head of R&D, Quadras Scientific Solutions
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2008-1877
Record Dates: First submitted 2019-10-24; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Intervention Model Description: Based on the log-transformed parameters, the following criteria were used to evaluate the bioequivalence between the test and reference products:
  * The 90% confidence interval of the relative mean AUCt of the test to reference products should be between80% and125%.
  * TherelativemeanCmaxofthetesttoreferenceproductsshouldbebetween80% and125%
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erlotinib HCl 150 mg (Experimental): Crossover
  Interventions: Drug: Erlotinib HCl 150 mg
- Tarceva® 150 mg (Active Comparator): Crossover
  Interventions: Drug: Tarceva®

INTERVENTIONS:
Drug: Erlotinib HCl 150 mg — Concentrations of erlotinib were measured from the samples collected over a 72 hour interval after receiving either Erotinib generic or Tarceva original. Later, after 14 days, a crossover was took place with the same measures.
  dosing in each period.
  Arms: Erlotinib HCl 150 mg
Drug: Tarceva® — Tarceva® 150 mg
  Arms: Tarceva® 150 mg

SUMMARY:
Theobjectiveofthisstudyistoevaluatethecomparativebioavailabilitybetween:

* ErlotinibHCl150mgTablets(Novopharm Limited,Canada)and
* Tarceva® 150mgTablets(Hoffmann-LaRocheLimited,Canada) afterasingle-doseinhealthysubjectsunderfastingconditions.

DETAILED DESCRIPTION:
This is a blinded,single-dose,randomized,two-period,two-sequence,two-treatment,cross over study, designed to evaluate the comparative bioavailability of two formulations of erlotinib HCl 150mg tablets administered to healthy male and female subjects under fasting conditions.

• SubjectswererandomlyassignedtooneofthetwodosingsequencesABorBA underfasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, post-menopausal and/or surgically sterile female subjects
* Healthy,non-smoking male subjects. Allsubjects willbe from 18 to 55 years ofage.

Exclusion Criteria:

* Known history or presence of any clinically significant medicalcondition.
* Known or suspected carcinoma.
* Presence ofclinically significant gastrointestinal disease or history of malabsorption within the last year.
* Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
* Use of tobacco or nicotine-containing products within 6 months priorto drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10-23 (Actual); Primary Completion 2008-11-09 (Actual); Study Completion 2008-11-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence (Biodisponibility) | 72 hours
  Compared Bioequivalence

IPD SHARING:
Plan to Share IPD: No